CLINICAL TRIAL: NCT01019746
Title: Comparison of Closed-oop of Propofol Versus Manual Control Using Bispectral Index (BIS)
Brief Title: Controlled Propofol Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: performance of a novel closed-loop propofol system, MUHC - Montreal General Hospitalization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN-07-002; GEN#07-002
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: HYPNOSIS
Keywords: Hypnosis with propofol
MeSH Terms: interventions — Propofol

ARMS (1):
- control propofol administration (Experimental)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — propofol administration

SUMMARY:
The purpose of this study is to compare the administration of the standard anesthetic agent (propofol) using this automatic system with the manual administration of propofol by the anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 90 years
* surgery lasting more than 30 min

Exclusion Criteria:

* inability to provide informed consent
* allergies to study drug

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Comparison of control administration of propofol with manual administration. | 1 year

SECONDARY OUTCOMES:
Emergence from anesthesia | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- MUHC - Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Hemmerling TM, Charabati S, Zaouter C, Minardi C, Mathieu PA. A randomized controlled trial demonstrates that a novel closed-loop propofol system performs better hypnosis control than manual administration. Can J Anaesth. 2010 Aug;57(8):725-35. doi: 10.1007/s12630-010-9335-z. Epub 2010 Jun 9. PMID 20533013